CLINICAL TRIAL: NCT07229170
Title: Changes in Taste Perception, Eating Habits, and Other Behavioral Aspects Associated With the Use of GLP-1 Receptor Agonists in Patients Undergoing Weight Loss Treatment: A Retrospective Observational Study.
Brief Title: Changes in Taste and Eating Habits Associated With GLP-1 Agonists in Weight Loss Patients
Acronym: GLP1-TASTE
Status: Not yet recruiting | Type: Observational
Sponsor: San Raffaele Telematic University (Other)
Responsible Party: Principal Investigator, Mauro Lombardo, Full professor in Human Nutrition, San Raffaele Telematic University
Other Study IDs: GLP1-TASTE
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Obesity & Overweight; Taste Alterations; Weight Loss; Eating Behavior Changes
Keywords: GLP-1 agonists; Obesity treatment; Weight loss; Taste perception; Eating habits; Observational study
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GLP-1 Agonist Treated Patients: This cohort includes adult patients aged 18-60 who have been treated with GLP-1 receptor agonists such as semaglutide or tirzepatide for weight loss in specialized nutrition centers in Italy. The study collects retrospective data on changes in taste perception, eating habits, body composition, and treatment adherence over a minimum duration of 12 weeks of therapy. No interventional treatments are administered as part of this observational study.

SUMMARY:
This observational retrospective study aims to evaluate changes in taste perception, eating habits, and behavioral aspects in adults treated with GLP-1 receptor agonists for weight loss. Participants include adults aged 18-60 receiving treatment at specialized nutrition centers in Italy. Data are collected from clinical records, dietary questionnaires, and metabolic assessments before and after at least 12 weeks of GLP-1 agonist treatment. The study's primary goal is to understand how these treatments affect food preferences and taste perception. Secondary outcomes include changes in body weight, body composition, gastrointestinal side effects, and treatment adherence. All data are anonymized and collected according to ethical guidelines.

DETAILED DESCRIPTION:
This retrospective observational study investigates changes in taste perception, eating habits, and other behavioral aspects associated with the use of GLP-1 receptor agonists in patients undergoing treatment for weight loss. The study includes adults aged 18-60 years who have been treated at specialized nutrition centers in Italy during 2025-2026. Data are collected retrospectively from clinical records, dietary questionnaires, bioimpedance analysis for body composition, and metabolic assessments conducted before and after at least 12 weeks of treatment with GLP-1 agonists such as semaglutide or tirzepatide.

The primary objective is to evaluate the impact of GLP-1 agonist treatment on food preferences and taste perception changes. Secondary objectives include quantifying changes in body weight, body mass index (BMI), and body composition (fat mass and lean mass), assessing gastrointestinal side effects, measuring total energy expenditure and physical activity variations, and estimating treatment adherence and discontinuation reasons.

Data collection involves anonymized extraction of demographic, anthropometric, clinical, dietary, and behavioral information in accordance with GDPR and ethical guidelines. The analysis is performed using statistical methods including paired t-tests, Wilcoxon tests, and regression models adjusted for age, sex, baseline BMI, diabetes status, and concomitant medications.

This study is non-profit and does not involve additional costs or interventions beyond routine clinical care. Ethical approval is pending and will be obtained before the study initiation. All procedures will comply with local regulations and ethical guidelines.

ELIGIBILITY:
Inclusion: Adults aged 18-60 years diagnosed with obesity and undergoing treatment with GLP-1 receptor agonists such as semaglutide or tirzepatide. Must have clinical records and dietary data available for at least 12 weeks of treatment.

Exclusion: Patients with conditions affecting taste independent of GLP-1 treatment, severe comorbidities, or inability to provide consent and data.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with obesity receiving GLP-1 agonist treatment at specialized nutrition centers in Italy, assessed retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in taste perception and food preferences | From baseline to 12 weeks after GLP-1 agonist treatment
  Assessment of patients' taste perception changes and shifts in eating habits using validated questionnaires and behavioral surveys.

SECONDARY OUTCOMES:
Change in body weight | From baseline to 12 weeks after treatment
  Measured in kilograms to assess weight loss effectiveness.
Gastrointestinal side effects | Throughout the treatment period
  Recording of nausea, vomiting, diarrhea, or other GI symptoms via patient reports.
Treatment adherence | Throughout the study duration
  Assessment of continued use and discontinuation reasons of GLP-1 agonists.

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Open University, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
At this time, there is no definitive plan to share individual participant data. Once the study is completed and data analysis finalized, decisions about data sharing will be made in accordance with institutional policies, ethical guidelines, and participant consent. If data sharing is pursued, de-identified datasets and supporting documents may be made available to qualified researchers upon reasonable request.

REFERENCES:
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185